CLINICAL TRIAL: NCT03696758
Title: Improving Right Ventricular Function in Young Adults Born Preterm: A Pilot Study
Brief Title: Improving Right Ventricular Function in Young Adults Born Preterm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0796; 1UL1TR002373-01 (NIH); A534285 (Other: UW Madison); SMPH/MEDICINE/PULMON MED (Other: UW Madison); Protocol Version 8/30/2018 (Other: UW Madison)
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Infant,Premature
Keywords: premature adults; premature; premature cardiac function; MRI; sildenafil; metoprolol; CMR
MeSH Terms: conditions — Premature Birth | interventions — Respiratory Physiological Phenomena; Metoprolol; Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Young adults born premature, recruited either from the National Lung Project Cohort or the general public, will undergo Cardiac Magnetic Resonance Imaging before and after medication administration. This will occur twice, on two separate visits. Subjects will be given sildenafil in between imaging scans at one visit, and will receive intravenous metoprolol in between scans at a separate visit. These visits can occur in either order. There will be a minimum period of 12 hours between drug interventions to ensure adequate drug wash-out.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil followed by Metoprolol (Experimental): Young adults born premature, recruited either from the National Lung Project Cohort or the general public, will undergo Cardiac Magnetic Resonance Imaging before and after medication administration. This will occur twice, on two separate visits. Subjects will be given sildenafil in between imaging scans at one visit, and will receive intravenous metoprolol in between scans at next visit. There will be a minimum period of 12 hours between drug interventions to ensure adequate drug wash-out. Subjects will also undergo pulmonary function testing and electrocardiogram.
  Interventions: Procedure: Pulmonary Function Testing; Procedure: Electrocardiogram; Procedure: Cardiac Magnetic Resonance Imaging; Drug: Metoprolol; Drug: Sildenafil
- Metoprolol followed by Sildenafil (Experimental): Young adults born premature, recruited either from the National Lung Project Cohort or the general public, will undergo Cardiac Magnetic Resonance Imaging before and after medication administration. This will occur twice, on two separate visits. Subjects will be given metoprolol in between imaging scans at one visit, and will receive intravenous sildenafil in between scans at next visit. There will be a minimum period of 12 hours between drug interventions to ensure adequate drug wash-out. Subjects will also undergo pulmonary function testing and electrocardiogram.
  Interventions: Procedure: Pulmonary Function Testing; Procedure: Electrocardiogram; Procedure: Cardiac Magnetic Resonance Imaging; Drug: Metoprolol; Drug: Sildenafil

INTERVENTIONS:
Procedure: Pulmonary Function Testing — Subjects will undergo spirometry, Plethysmography, and diffusion capacity.
Procedure: Electrocardiogram — Subjects will undergo an electrocardiogram to ensure sinus rhythm
Procedure: Cardiac Magnetic Resonance Imaging — Subjects will undergo positron magnetic resonance imaging to detect images of the heart
Drug: Metoprolol — Subjects will receive intravenous metoprolol. Dose titrated 1-5 mg every 2 minutes to achieve goal heart rate of 55-65 beats per minute, or for subjects with a resting heart rate already at goal, titrated to achieve a 10-15% reduction in heart rate.
  Other Names: Lopressor; Metolar XR
Drug: Sildenafil — Subjects will receive a 50 milligram tablet of sildenafil (to be taken orally)
  Other Names: Revatio

SUMMARY:
The purpose of this research is to evaluate the short-term effects of sildenafil and metoprolol on heart function in young adults born premature.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the short-term therapeutic effects of sildenafil and metoprolol on right ventricular function in young adults born premature using novel 4-Dimensional flow Cardiac Magnetic Resonance Imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Male or female aged 18-35
3. History of preterm birth (either a or b):

   1. Participant in the Newborn Lung Project (birth year 1988-1991, birth weight <1500 g)
   2. Non-NLP participant, with birth weight <1500 g and gestational age 32 weeks or less, verified by medical records

Exclusion Criteria:

1. Pregnant or lactating
2. Use of prescribed medications that would interfere with study medications

   1. Sildenafil: Use of phosphodiesterase type 5 inhibitors (sildenafil, tadalafil, vardenafil), nitrates, soluble guanylate cyclase inhibitor (riociguat) within 48 hours of study visit
   2. Metoprolol: Use of nodal blocking agents including beta blockers, non-dihydropyridine calcium channel blockers (i.e. diltiazem), and anti-arrhythmics (i.e. amiodarone)
3. Presence of known comorbidities for which these therapeutic interventions would be contraindicated:

   1. Moderate to severe heart failure
   2. Severe bradycardia (heart rate <45), or second or third-degree heart block
   3. Systolic blood pressure <90 mmHg or >190 mmHg
   4. Angina
   5. Severe peripheral arterial circulatory disorders
   6. History of severe bronchospasm
4. Presence of any implanted device incompatible with CMR imaging
5. Known allergic or hypersensitivity reaction to components of the study medications
6. Any other reason for which the investigator deems a subject unsafe or inappropriate for study participation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara N Goss, MD, Principal Investigator — University of Wisconsin-Madison School of Medicine and Public Health
Locations (1):
- University of Wisconsin-Madison School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to COVID shut down, 1 participant was excluded from the study before assignment to groups
Period: First Intervention
Arm/Group | Sildenafil Followed by Metoprolol | Metoprolol Followed by Sildenafil
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0
Period: Wash Out>12 Hours
Arm/Group | Sildenafil Followed by Metoprolol | Metoprolol Followed by Sildenafil
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Sildenafil Followed by Metoprolol | Metoprolol Followed by Sildenafil
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Young Adults Born Premature: Young adults born premature, recruited either from the National Lung Project Cohort or the general public, will undergo Cardiac Magnetic Resonance Imaging before and after medication administration. This will occur twice, on two separate visits. Subjects will be given sildenafil in between imaging scans at one visit, and will receive intravenous metoprolol in between scans at a separate visit. These visits can occur in either order. Subjects will also undergo pulmonary function testing and electrocardiogram.
  Pulmonary Function Testing: Subjects will undergo spirometry, Plethysmography, and diffusion capacity.
  Electrocardiogram: Subjects will undergo an electrocardiogram to ensure sinus rhythm Cardiac Magnetic Resonance Imaging: Subjects will undergo positron magnetic resonance imaging to detect images of the heart Metoprolol: Subjects will receive intravenous metoprolol Sildenafil: Subjects will receive a 50 milligram tablet of sildenafil (to be taken orally)
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.8 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Gestational age (Neonatal Characteristics) [Mean (Standard Deviation); unit: Weeks] | 28.9 (2.7)
Birth weight (Neonatal Characteristics) [Mean (Standard Deviation); unit: gram] | 1116 (342)

OUTCOME MEASURES:

1. Primary Outcome: Right Ventricular Energetic Efficiency Pre and Post Metoprolol
Description: To characterize energy efficiency, the total Kinetic Energy across the cardiac cycle is normalized to right ventricular end-diastolic volume and left ventricular end-diastolic volume, respectively. Analysis will be completed in blinded fashion. Two imaging scans will be done - one pre and one post Metoprolol intervention. Total time from Pre-intervention scan till post intervention scan may take up to 2 hours.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: µJ/ml
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
µJ/ml
  Pre Metoprolol | 15.5 (2.6)
  Post Metoprolol | 12.7 (2.5)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.004, Wilcoxon Signed Rank Test — p value is 0.004 for 'Pre-Metoprolol' vs 'post-Metoprolol' subgroup

2. Primary Outcome: Right Ventricular Energetic Efficiency Pre and Post Sildenafil
Description: To characterize energy efficiency, the total Kinetic Energy across the cardiac cycle is normalized to right ventricular end-diastolic volume and left ventricular end-diastolic volume, respectively. Analysis will be completed in blinded fashion. Two imaging scans will be done - one pre and one post Sildenafil intervention. Total time from Pre-intervention scan till post intervention scan may take up to 2 hours.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: µJ/ml
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
µJ/ml
  Pre-Sildenafil | 15.8 (3.7)
  Post-Sildenafil | 17.9 (6.2)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.13, Wilcoxon Signed Rank Test — P-Value is 0.13 for 'Pre-Sildenafil' vs 'Post-Sildenafil' subgroup

3. Secondary Outcome: Left Ventricular Energetic Efficiency Pre and Post Metoprolol
Description: Kinetic energy (from 4D flow) normalized to ventricular volume (from MRI). Participants will receive intravenous metoprolol in between scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: µJ/ml
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
µJ/ml
  Pre-Metoprolol | 11.6 (5)
  Post-Metoprolol | 9.5 (3.7)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — descriptive statistics; p = 0.004, Wilcoxon Signed Rank Test — p value is 0.004 for 'Pre-Metoprolol' vs 'post-Metoprolol' subgroup

4. Secondary Outcome: Right Ventricular Ejection Fraction Pre and Post Metoprolol
Description: Participants will receive intravenous metoprolol in between scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
percentage
  Pre-Metoprolol | 55 (8)
  Post-Metoprolol | 51 (8)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.1, Wilcoxon Signed Rank Test — p value is 0.10 for 'Pre-Metoprolol' vs 'post-Metoprolol' subgroup

5. Secondary Outcome: Right Ventricular Stroke Volume Pre and Post Metoprolol
Description: Participants will receive intravenous metoprolol in between scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Metoprolol | 41.5 (7.6)
  Post-Metoprolol | 37.7 (5.1)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.09, Wilcoxon Signed Rank Test — p value is 0.09 for 'Pre-Metoprolol' vs 'post-Metoprolol' subgroup

6. Secondary Outcome: Right Ventricular Systolic Volume Pre and Post Metoprolol
Description: Participants will receive intravenous metoprolol in between scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Metoprolol | 33.7 (7.5)
  Post-Metoprolol | 36.6 (9.3)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.10, Wilcoxon Signed Rank Test — p value is 0.10 for 'Pre-Metoprolol' vs 'post-Metoprolol' subgroup

7. Secondary Outcome: Right Ventricular Diastolic Volume Pre and Post Metoprolol
Description: Participants will receive intravenous metoprolol in between scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Metoprolol | 75.2 (9.8)
  Post-Metoprolol | 74.4 (9.4)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.82, Wilcoxon Signed Rank Test — p value is 0.82 for 'Pre-Metoprolol' vs 'post-Metoprolol' subgroup

8. Secondary Outcome: Left Ventricular Ejection Fraction Pre and Post Metoprolol
Description: Participants will receive intravenous metoprolol in between scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
percentage
  Pre-Metoprolol | 60 (6)
  Post-Metoprolol | 58 (8)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.30, Wilcoxon Signed Rank Test — p value is 0.30 for 'Pre-Metoprolol' vs 'post-Metoprolol' subgroup

9. Secondary Outcome: Left Ventricular Stroke Volume Pre and Post Metoprolol
Description: Participants will receive intravenous metoprolol in between scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Metoprolol | 43.7 (7.1)
  Post-Metoprolol | 41.4 (5.6)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.36, Wilcoxon Signed Rank Test — p value is 0.36 for 'Pre-Metoprolol' vs 'post-Metoprolol' subgroup

10. Secondary Outcome: Left Ventricular Systolic Volume Pre and Post Metoprolol
Description: Participants will receive intravenous metoprolol in between scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Metoprolol | 28.8 (6)
  Post-Metoprolol | 30.6 (8.2)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.36, Wilcoxon Signed Rank Test — p value is 0.36 for 'Pre-Metoprolol' vs 'post-Metoprolol' subgroup

11. Secondary Outcome: Left Ventricular Diastolic Volume Pre and Post Metoprolol
Description: Participants will receive intravenous metoprolol in between scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Metoprolol | 72.5 (10.1)
  Post-Metoprolol | 72.1 (9.7)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.65, Wilcoxon Signed Rank Test — P-Value is 0.65 for 'Pre-Metoprolol' vs 'post-Metoprolol' subgroup

12. Secondary Outcome: Left Ventricular Energetic Efficiency Pre and Post Sildenafil
Description: Kinetic energy (from 4D flow) normalized to ventricular volume (from MRI). Participants will be given sildenafil in between imaging scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: µJ/ml
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
µJ/ml
  Pre-Sildenafil | 11.1 (2.8)
  Post-Sildenafil | 12.3 (4)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.25, Wilcoxon Signed Rank Test — P-Value is 0.25 for 'Pre-Sildenafil' vs 'Post-Sildenafil' subgroup

13. Secondary Outcome: Right Ventricular Ejection Fraction Pre and Post Sildenafil
Description: Participants will be given sildenafil in between imaging scans. The term "ejection fraction" refers to the percentage of blood that's pumped out of a filled ventricle with each heartbeat.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
percentage
  Pre-Sildenafil | 53 (7)
  Post-Sildenafil | 55 (10)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.43, Wilcoxon Signed Rank Test — P-Value is 0.43 for 'Pre-Sildenafil' vs 'Post-Sildenafil' subgroup

14. Secondary Outcome: Right Ventricular Stroke Volume Pre and Post Sildenafil
Description: Participants will be given sildenafil in between imaging scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Sildenafil | 40.4 (5.3)
  Post-Sildenafil | 41.3 (10.7)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.66, Wilcoxon Signed Rank Test — P-Value is 0.66 for 'Pre-Sildenafil' vs 'Post-Sildenafil' subgroup

15. Secondary Outcome: Right Ventricular Systolic Volume Pre and Post Sildenafil
Description: Participants will be given sildenafil in between imaging scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Sildenafil | 35.8 (8.5)
  Post-Sildenafil | 33.3 (7.3)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.13, Wilcoxon Signed Rank Test — P-Value is 0.13 for 'Pre-Sildenafil' vs 'Post-Sildenafil' subgroup

16. Secondary Outcome: Right Ventricular Diastolic Volume Pre and Post Sildenafil
Description: Participants will be given sildenafil in between imaging scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Sildenafil | 76.2 (9.1)
  Post-Sildenafil | 74.6 (11.3)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.57, Wilcoxon Signed Rank Test — P-Value is 0.57 for 'Pre-Sildenafil' vs 'Post-Sildenafil' subgroup

17. Secondary Outcome: Left Ventricular Ejection Fraction Pre and Post Sildenafil
Description: Participants will be given sildenafil in between imaging scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
percentage
  Pre-Sildenafil | 60 (7)
  Post-Sildenafil | 63 (8)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.25, Wilcoxon Signed Rank Test — P-Value is 0.25 for 'Pre-Sildenafil' vs 'Post-Sildenafil' subgroup

18. Secondary Outcome: Left Ventricular Stroke Volume Pre and Post Sildenafil
Description: Participants will be given sildenafil in between imaging scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Sildenafil | 43.1 (8.1)
  Post-Sildenafil | 45.7 (9.2)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.07, Wilcoxon Signed Rank Test — P-Value is 0.07 for 'Pre-Sildenafil' vs 'Post-Sildenafil' subgroup

19. Secondary Outcome: Left Ventricular Systolic Volume Pre and Post Sildenafil
Description: Participants will be given sildenafil in between imaging scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Sildenafil | 28.1 (5.4)
  Post-Sildenafil | 26.6 (5.7)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.36, Wilcoxon Signed Rank Test — P-Value is 0.36 for 'Pre-Sildenafil' vs 'Post-Sildenafil' subgroup

20. Secondary Outcome: Left Ventricular Diastolic Volume Pre and Post Sildenafil
Description: Participants will be given sildenafil in between imaging scans.
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Young Adults Born Premature
Number analyzed (Participants) | 9
ml/m^2
  Pre-Sildenafil | 71.2 (8.8)
  Post-Sildenafil | 72.2 (8.0)
Statistical Analysis 1: Comparison: Young Adults Born Premature; Test type: Other — Descriptive statistics; p = 0.91, Wilcoxon Signed Rank Test — P-Value is 0.91 for 'Pre-Sildenafil' vs 'Post-Sildenafil' subgroup

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Sildenafil Followed by Metoprolol: Young adults born premature, recruited either from the National Lung Project Cohort or the general public, will undergo Cardiac Magnetic Resonance Imaging before and after medication administration. This will occur twice, on two separate visits. Subjects will be given sildenafil in between imaging scans at one visit, and will receive intravenous metoprolol in between scans at next visit. There will be a minimum period of 12 hours between drug interventions to ensure adequate drug wash-out. Subjects will also undergo pulmonary function testing and electrocardiogram.
  Pulmonary Function Testing: Subjects will undergo spirometry, Plethysmography, and diffusion capacity.
  Electrocardiogram: Subjects will undergo an electrocardiogram to ensure sinus rhythm
  Cardiac Magnetic Resonance Imaging: Subjects will undergo positron magnetic resonance imaging to detect images of the heart
  Metoprolol: Subjects will receive intravenous metoprolol
  Sildenafil: Subjects will receive a 50 milligram tablet of sildenafil (to be taken orally)
Arm/Group | Sildenafil Followed by Metoprolol | Metoprolol Followed by Sildenafil
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT03696758/Prot_SAP_000.pdf